CLINICAL TRIAL: NCT03653156
Title: China Cognition and Aging Study: a Multi-center, National-wide, Longitudinal Study in China
Brief Title: China Cognition and Aging Study
Acronym: COAST
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Chao Yang Hospital (Other); Fu Xing Hospital, Capital Medical University (Other); Peking Union Medical College Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Chinese PLA General Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Geriatric Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Fujian Medical University Union Hospital (Other); Guangzhou Psychiatric Hospital (Other Government); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Handan Central Hospital (Other); Hebei General Hospital (Other); First Hospital of Shijiazhuang City (Other); Tangshan Worker's Hospital (Other); Hunan Provincial People's Hospital (Other); Kaifeng Central Hospital (Other); People's Hospital of Zhengzhou University (Other); Zhongnan Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Tongji Hospital (Other); People's Hospital Affiliated Hubei Medical University (Unknown); The Third Xiangya Hospital of Central South University (Other); Xiangya Hospital of Central South University (Other); The First Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other); Subei People's Hospital of Jiangsu (Unknown); Nantong University Affiliated Hospital (Unknown); Mineral General Hospital, Xuzhou (Unknown); Jiangxi Provincial People's Hopital (Other); Anshan Central Hospital (Other); Affiliated Zhongshan Hospital of Dalian University (Other); First Hospital of China Medical University (Other); Baotou Central Hospital (Other); General Hospital of Ningxia Medical University (Other); The People's Hospital of Ningxia (Other); The Affiliated Hospital of Qingdao University (Other); The 960th Hospital of PLA (Unknown); Qilu Hospital of Shandong University (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Shandong Provincial Hospital (Other Government); Qingdao Municipal Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Tang-Du Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Ruijin Hospital (Other); RenJi Hospital (Other); Shanghai Changzheng Hospital (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Tianjin Huanhu Hospital (Other); Tianjin Medical University General Hospital (Other); Traditional Chinese Medicine Hospital of Xinjiang Autonomous Region (Unknown); Ningbo Medical Center Lihuili Hospital (Other Government); First Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); Shao Yifu Hospital of Zhejiang Medical University (Unknown); Zhejiang Provincial People's Hospital (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); People's Hospital of Chongqing (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other); Zigong No.1 Peoples Hospital (Other)
Responsible Party: Principal Investigator, Jianping Jia, Chief Director, Capital Medical University
Other Study IDs: SYXWJ001
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Mild Cognitive Impairment(MCI); Alzheimer Disease, Late Onset; Familial Alzheimer Disease (FAD); Vascular Dementia (VaD); Normal Control; Non-Alzheimer Degenerative Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Plasma, CSF, saliva and biopsy and autopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Mild cognitive impairment (MCI) and its subtypes: MCI cohort consists of mild cognitive impairment subjects with memory loss as predominant symptom, including amnestic mild cognitive impairment and vascular cognitive impairment no dementia, which recruit from community population and hospital population.
- Sporadic Alzheimer's disease (SAD): SAD cohort consists of mild to moderate sporadic Alzheimer's disease subjects, which recruit from community population and hospital population.
- Familial Alzheimer's disease (FAD): FAD cohort consists of familial Alzheimer disease subjects with known or unknown mutations, which recruit from community population and hospital population.
- Vascular dementia(VaD）: VaD cohort consists of cognitive impairment subjects caused by cerebral vessel disease, including vascular dementia and mixes dementia, which recruit from community population and hospital population.
- Normal control: Normal control cohort consists of cognitive normal subjects with ApoE ε4 positive or negative, which recruit from community population and hospital population.
- Non-Alzheimer degenerative dementia: Frontotemporal dementia (FTD); or Parkinson's disease dementia (PDD); or dementia with Lewy bodies (DLB); or corticobasal degeneration (CBD); or dementia not otherwise specified.

SUMMARY:
The aim of this study is to establish and perfect the China Cognition and Aging Study (China COAST) cohort, to clarify the epidemiology, influencing factors, genetic characteristics, pathogenesis, disease characteristics and diagnosis and treatment status of dementia and its subtypes in China. It is of great significance to establish a relatively comprehensive national database of cognitive disorders, improve the clinical diagnosis and treatment level of cognitive disorders, and formulate prevention and treatment strategies for dementia. The primary aims of China COAST are as follows:

1. To use the prospective cohort to establish a large database research platform, so as to provide comprehensive epidemiological data, clinical and neuropsychological evaluation data, biological samples, and laboratory tests and imaging data.
2. To update the prevalence and incidence rate of dementia and its subtypes every 2-3 years, and clarify the conversion pattern from normal elderly to MCI and from MCI to dementia.
3. To explore the known or unknown protective and risk factors of dementia and its major subtypes (AD, VaD, other dementia).
4. To discover new pathogenic genes and susceptible genes of dementia and its major subtypes (AD and VaD), as well as new mutation sites of known pathogenic genes. To study the genetic variation, mutation and polymorphism of PSEN1, PSEN2, APP and APOE genes in dementia patients, and to understand their distribution and roles in the pathogenesis.
5. To study the biomarkers (body fluid, genetics, imaging) with diagnostic value of MCI, AD (sporadic and familial) and VaD, to define their cut-off values, and to establish prediction models.
6. To study the diagnostic criteria of cognitive normal, MCI, dementia and their subtypes (clinical and molecular subtypes) in the cohort, and to make psychological assessment scales with high sensitivity and specificity, and in line with the characteristics of Chinese people.
7. To find potentially modifiable risk factors for dementia and to study the prevention and intervention effect of non-pharmacological treatment on APOE ε4 carriers, MCI and AD or other dementia patients，which included improvements in education, nutrition, health care, and lifestyle changes. This needs a long time follow-up.
8. To explore the relationship between dementia as well as its major subtype AD and cerebral and systemetic circulatory disorders (for example, mixed dmentia), as well as potential therapeutic strategies.
9. To carry out investigation and researches about dementia related education, improve the awareness of dementia, and strengthen the management of dementia.
10. To investigate the level of stigma and discrimination and its influencing factors in patients with Alzheimer's disease and their caregivers.

DETAILED DESCRIPTION:
This study involved participants including Mild cognitive impairment (MCI) and its subtypes、Sporadic Alzheimer's disease (SAD)、 Familial Alzheimer's disease (FAD)、Vascular dementia (VaD)、Normal control in community population and hospital population. Research contents are as follow:

1. Through the collection of basic demographic information and clinical data from the multi-center cohort, we will calculate the prevalence and incidence rate of AD, VaD, other dementia (mixed dementia, FTD, DLB, PDD, alcohol dementia, hydrocephalus dementia, post-traumatic dementia, etc.), and update the numbers every 1-2 years.
2. To clarify the conversion pattern from normal elderly to MCI and from MCI to dementia. Through the collection and analysis of current medical history, past history, family history, living habits, drug use, physical examination and other information, we will explore the protective and risk factors of dementia and its main subtypes (AD, VaD, Other dementia), including age, gender, education level, rural/urban, marital status, parental dementia history, dietary habbit, blood pressure, drinking, smoking, diabetes, hyperlipidemia, cerebrovascular disease, heart disease, depression, hearing impairment, exercise habits (Tai chi, etc.), dementia specialist influence on patients, occupation, BMI, lifestyle changes, air pollution, head injury , social contact, low-income, and other unknown protective or risk factors. To investigate the role of ApoE gene, especially ApoEε4 in the disease onset and development, and to explore the non-pharmacological interventions For the study purpose we do follow-up every 2or 3 years.
3. By using exome sequencing, GWAS, WGS and other methods, we will search for new mutations of known pathogenic genes (APP, PSEN1, PSEN2) of AD in China, find new pathogenic genes and susceptible genes of dementia and its main subtypes (AD and VaD), and understand their distribution. We will explore the independent and combined effect of susceptibility gene variation on the risk of illness in Chinese AD population, and to obtain the key mutation sites that have a clear relationship with the incidence of AD. We will do regular follow up visits for the FAD members with new mutations of pathogenic genes, and clarify the important role of new mutations of pathogenic genes during the onset and progression of AD.
4. We will collect the biofluids (blood, cerebrospinal fluid, urine, etc.) and 18F-FDG / 11C-PIB PET/MR multimodal imaging data from people with normal cognition, MCI, AD (sporadic and familial) and VaD, and conduct regular follow up. Discover and verify the SAD related susceptible gene and FAD related pathogenic gene mutation. Through analyzing the imaging data (such as MRI brain regional volume, 18F-FDG PET and cortical Aβ load), cerebrospinal fluid and plasma markers (such as Aβ, T-tau and P-tau) and clinical features (such as psychiatric symptoms and age of onset), we will develop gene chip with high sensitivity and high specificity for early screening of dementia; develop diagnostic kits for biofluid markers (blood and cerebrospinal fluid); determine imaging cut-off values at all stages of dementia in Chinese people. We will do correlation analysis to establish early diagnosis and risk prediction model for dementia, and verify the newly developed instruments that can detect the peripheral markers of dementia patients and predict the disease progression in national large sample.
5. Through the unified and standardized neuropsychological scales, including MMSE, MoCA, CDR, NPI, ADL, etc, we will conduct investigation to subjects in baseline and follow-up period, and analyze the changes of cognitive function, ability of daily life and mental behavior symptoms in different cognitive disorders. According to the social, cultural and material changes in China in recent years, we will develop psychological assessment scales with high sensitivity and specificity, and in line with the characteristics of Chinese people. Meanwhile, on the basis of the international diagnostic standards of various subtypes of dementia, combined with the etiology, clinical manifestations, scale classification, imaging characteristics, biofluid examination, etc., we will study the novel typing method and diagnostic standards of cognitive normal, MCI, dementia and its subtypes (clinical and molecular subtypes) in Chinese population.
6. Through designing randomized controlled trials, we will study the systematic and effective NPT intervention program, including lifestyle (diet and sleep habits, smoking, drinking and social networking), health products, exercise habits, cognitive training, risk factor control, etc. We will explore the quantitative and objective evaluation criteria of NPT in AD and dementia, clarify its prevention and control efficacy on APOE ε4 carriers, MCI and dementia patients, and potential neurobiological mechanism. At the same time, we will carry out dementia related education in the community, improve the public knowledge, attention and awareness of dementia, so that patients can get early detection, early diagnosis and early intervention.
7. To explore the relationship between dementia as well as its major subtype AD and cerebral circulatory disorders (cerebral ischemic and hemorrhage diseases, cerebral arteriosclerosis and stenosis, cerebral venous diseases, etc.), especially clarify the relationship between chronic cerebral ischemia and AD, as well as its effect on AD onset, and whether or not it's risk factor for AD. Whether the therapeutic strategies for cerebral circulatory disorders should be included in the treatment of AD.

ELIGIBILITY:
Community population: age ≥ 55 years, male or female, with consent to participant the study.

Hospital population: subjects are all over 18 years old. Through clinical evaluation, neuropsychological test, imaging examination, blood and cerebrospinal fluid examination, etc, we will comprehensively evaluate the cognitive function and various test measures.

(1) MCI and its subtypes

Inclusion criteria:

1. Diagnosis according to 2004 Peterson's MCI criteria.
2. CDR = 0.5.
3. Memory loss is prominent, and may also be with other cognitive domain dysfunction.
4. Insidious onset, slow progress.
5. Not reaching the level of dementia.

Exclusion criteria:

1. With history of stroke and a neurological focal sign, the imaging findings are consistent with cerebral small vessal disease (Fazekas score ≥ 2 points).
2. Other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.).
3. Other systemic diseases that can cause cognitive impairment (such as liver, renal and thyroid insufficiency, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.).
4. Mental and neurodevelopmental retardation.
5. Contraindications to MRI.
6. Suffering from a disease that cannot be combined with cognitive examination.
7. Refuse to draw blood.
8. Refuse to sign the informed consent at baseline

(2) Sporadic Alzheimer's disease (SAD)

Inclusion criteria:

1. Dementia is diagnosed according to the criteria described by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-R). The diagnosis of AD is made using the National Institute of Neurologic and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) or National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria.
2. Subjects and their informed persons can complete relevant and follow- up examinations.
3. Subjects or their authorized legal guardians sign the informed consent.

Exclusion criteria:

1. With a family history of dementia.
2. Other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.).
3. Other systemic diseases that can cause cognitive impairment (such as liver, renal and thyroid insufficiency, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.).
4. Mental and neurodevelopmental retardation.
5. Contraindications to MRI.
6. Suffering from a disease that cannot be combined with cognitive examination.
7. Refuse to draw blood.
8. Refuse to sign the informed consent at baseline

(3) Familial Alzheimer's disease (FAD)

Inclusion criteria:

1. Written informed consent obtained from participant or legal guardian prior to any study-related procedures.
2. Members in FAD pedigree (FAD is defined as at least two first- degree relatives suffer from AD).
3. Aged 18 (inclusive) or older.
4. At least two persons who can provide reliable information for the study. Note: Dementia is diagnosed according to the criteria described by DSM-IV-R. The diagnosis of AD is made using NINCDS-ADRDA or NIA-AA criteria. A diagnosis of MCI is assigned according to Petersen criteria.

Exclusion criteria:

1. Dementia caused by other factors such as depression, other psychiatric illnesses, thyroid dysfunction, encephalitis, multiple sclerosis, brain trauma, brain tumor, syphilis, acquired immunodeficiency syndrome (AIDS), Creutzfeldt-Jakob disease and other types of dementias such as vascular dementia (VaD), frontotemporal dementia (FTD), dementia with Lewy bodies (DLB), and Parkinson's disease dementia (PDD).
2. MRI and laboratory tests do not support or rule out a diagnosis of AD.
3. Severe circulatory, respiratory, urinary, digestive, hematopoietic diseases (such as unstable angina, uncontrollable asthma, active gastric bleeding) and cancer.
4. Participant has severe psychiatric illness or severe dementia that would interfere in completing initial and follow-up clinical assessments.
5. With history of alcohol or drug abuse.
6. Pregnant or lactating women.
7. No reliable insiders.
8. Refuse to sign the informed consent at baseline.

(4) Vascular dementia (VaD)

Inclusion criteria:

Diagnosis for probable VaD according to NINDS-AIREN diagnostic criteria.

MRI inclusion criteria:

All patients who meet clinical inclusion criteria should accept MRI scans which include an assessment of hippocampal volume.

1. multiple (≥3) supratentorial subcortical small infarcts (3-20 mm in diameter) with or without any degree of white matter lesion (WML); or moderate to severe WML (Fazekas score ≥ 2), with or without small infarction; or ≥ 1 subcortical small infarct in key regions, such as caudate nucleus, globus pallidus, or thalamus.
2. no cortical and watershed infarction, hemorrhage, hydrocephalus, or WML with specific causes (such as multiple sclerosis).
3. no hippocampus or entorhinal cortex atrophy (MTA score = 0 point).

Exclusion criteria:

1. Other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.).
2. Other systemic diseases that can cause cognitive impairment (such as liver insufficiency, renal insufficiency, thyroid insufficiency, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.).
3. With a history of mental illness or those with congenital mental retardation.
4. Suffering from a disease that cannot be combined with a cognitive examination.
5. Contraindications to MRI.
6. Refuse to draw blood.
7. Refuse to sign informed consent.

(5) Normal control

Inclusion criteria:

1. Aged 18 (inclusive) or above.
2. Normal MMSE and MoCA evaluations. MMSE>19 points for illiteracy, >24 points for those educated less than 7 years, >27 points for those educated equal to or more than 7 years. MoCA>13 points for illiteracy, >19 points for those educated less than 7 years, >24 points for those educated equal to or more than 7 years.

Exclusion criteria:

1. Subjects with abnormal MMSE or MoCA scores.
2. Subjects with a history of cerebral infarction, traumatic brain injury or related manifestations in MRI.
3. Other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.).
4. Other systemic diseases that can cause cognitive impairment (such as liver, renal and thyroid insufficiency, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.).
5. Mental and neurodevelopmental retardation.
6. Suffering from a disease that cannot be combined with a cognitive examination.
7. Contraindications to MRI.
8. Refuse to draw blood.
9. Refuse to sign the informed consent at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mild cognitive impairment (MCI) and its subtypes、Sporadic Alzheimer's disease (SAD)、 Familial Alzheimer's disease (FAD)、Vascular dementia (VaD)、Normal control in Community population and Hospital population.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2038-01-01 (Estimated); Study Completion 2038-01-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of MCI and AD measured using a population-based cross-sectional survey with a multistage cluster sampling design | an average of 2 years
The conversion rate of normal to MCI to AD in Chinese | an average of 2 years
The biomarkers for normal (pre-MCI), MCI and AD diagnosis | an average of 2 years
  Humoral biomarkers are included Aβ42, Aβ40, phosphated tau and total tau in plasma, cerebrospinal fluid, saliva, and urine. Imaging biomarkers are included cerebral volume, glucose metabolism, amyloid and tau deposition of whole brain or hippocampus.
The risk factors (genetic and environmental factors) for MCI, AD and VCI at genomic and expression levels | an average of 2 years
  Discover risk factors including genetic susceptibility loci (APOE genes and other risk genes) using gene sequencing, cardiovascular risk factors (blood glucose, cholesterol, homocysteine) using laboratory tests, and unhealthy lifestyle using questionnaire.
The effective non-pharmacologic treatment(NPT) intervention | an average of 2 years
  The effective non-pharmacologic treatment(NPT) intervention- including lifestyle(diet and sleep habits, smoking, drinking and social networking), health products, exercise habits, cognitive training, risk factor control- on APOE ε4 carriers, MCI and dementia patients using questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, Doctor, Study Chair — Xuanwu Hospital of Capital Medical University
Locations (65):
- China (65):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Geriatric Hospital, Changping, Beijing Municipality
  - Beijing Chao Yang Hospital, Chaoyang, Beijing Municipality
  - China-Japan Friendship Hospital, Chaoyang, Beijing Municipality
  - Dongfang Hospital Affiliated to Beijing University of Chinese Medicine, Fengtai, Beijing Municipality
  - Chinese PLA General Hospital, Haidian, Beijing Municipality
  - Fu Xing Hospital, Capital Medical University, Haidian, Beijing Municipality
  - Peking University Third Hospital, Haidian, Beijing Municipality
  - Peking Union Medical College Hospital, Xicheng, Beijing Municipality
  - Peking University First Hospital, Xicheng, Beijing Municipality
  - Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Yuzhong, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Yuzhong, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fujian, Guangdong
  - Guangzhou Psychiatric Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Zhongshan, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital Of Guizhou Medical University, Guiyang, Guizhou
  - Handan Central Hospital, Handan, Hebei
  - First Hospital of Shijiazhuang City, Shijiazhuang, Hebei
  - Tangshan Worker's Hospital, Tangshan, Hebei
  - Hebei General Hospital, Zhijiazhuang, Hebei
  - First Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - People's Hospital Affiliated Hubei Medical University, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Wuhan, Hunan
  - Wuhan University Zhongnan Hospital, Wuhan, Hunan
  - Xiangya Hospital of Central South University, Wuhan, Hunan
  - Nantong University Affiliated Hospital, Nantong, Jiangsu
  - Subei People's Hospital of Jiangsu, Subei, Jiangsu
  - Mineral General Hospital, Xuzhou, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - China-Japan friendship Hospital of Jilin university, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Changda Hospital, Anshan, Anshan, Liaoning
  - Affiliated Zhongshan hospital of Dalian university, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - First Hospital of China Medical University, Shenyang, Liaoning
  - Baotou Central Hospital, Baotou, Nei Monggol
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The People's Hospital of Ningxia, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jining, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao, Shandong
  - QingDao Municipal Hospital, Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The 88th Hospital of PLA, Tai’an, Shandong
  - Shanghai Changzheng Hospital, Huangpu, Shanghai Municipality
  - Ruijin Hospital, Luwan, Shanghai Municipality
  - RenJi Hospital, Putong, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - First Affiliated Hospital Xi'an Jiaotong University, Xi’an, Shanxi
  - Tang-Du Hospital, Xi’an, Shanxi
  - Afﬁliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Zigong First People's Hospital, Zigong, Sichuan
  - Tianjin Huanhu Hospital, Xianshuigu, Tianjin Municipality
  - Tianjin Medical University General Hospital, Xiaobailou, Tianjin Municipality
  - Traditional Chinese Medicine Hospital of Xinjiang Autonomous Region, Ürümqi, Xinjiang
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Shao Yifu Hospital of Zhejiang Medical University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo City Medical Treatment Center Lihuili Hospital, Ningbo, Zhejiang
  - First Affiliated Hospital of Wenzhou Medical Univeristy, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhou A, Jia J. A screen for cognitive assessments for patients with vascular cognitive impairment no dementia. Int J Geriatr Psychiatry. 2009 Dec;24(12):1352-7. doi: 10.1002/gps.2265. PMID 19347838
- [Result] Zhou A, Jia J. Different cognitive profiles between mild cognitive impairment due to cerebral small vessel disease and mild cognitive impairment of Alzheimer's disease origin. J Int Neuropsychol Soc. 2009 Nov;15(6):898-905. doi: 10.1017/S1355617709990816. PMID 19891819
- [Result] Bai F, Liao W, Watson DR, Shi Y, Yuan Y, Cohen AD, Xie C, Wang Y, Yue C, Teng Y, Wu D, Jia J, Zhang Z. Mapping the altered patterns of cerebellar resting-state function in longitudinal amnestic mild cognitive impairment patients. J Alzheimers Dis. 2011;23(1):87-99. doi: 10.3233/JAD-2010-101533. PMID 20930266
- [Result] Han Y, Wang J, Zhao Z, Min B, Lu J, Li K, He Y, Jia J. Frequency-dependent changes in the amplitude of low-frequency fluctuations in amnestic mild cognitive impairment: a resting-state fMRI study. Neuroimage. 2011 Mar 1;55(1):287-95. doi: 10.1016/j.neuroimage.2010.11.059. Epub 2010 Nov 28. PMID 21118724
- [Result] Lu J, Li D, Li F, Zhou A, Wang F, Zuo X, Jia XF, Song H, Jia J. Montreal cognitive assessment in detecting cognitive impairment in Chinese elderly individuals: a population-based study. J Geriatr Psychiatry Neurol. 2011 Dec;24(4):184-90. doi: 10.1177/0891988711422528. PMID 22228824
- [Result] Shi FD, Jia JP. Neurology and neurologic practice in China. Neurology. 2011 Nov 29;77(22):1986-92. doi: 10.1212/WNL.0b013e31823a0ed3. PMID 22123780
- [Result] Han Y, Jia J, Jia XF, Qin W, Wang S. Combination of plasma biomarkers and clinical data for the detection of sporadic Alzheimer's disease. Neurosci Lett. 2012 May 16;516(2):232-6. doi: 10.1016/j.neulet.2012.03.094. Epub 2012 Apr 7. PMID 22503901
- [Result] Li F, Jia XF, Jia J. The Informant Questionnaire on Cognitive Decline in the Elderly individuals in screening mild cognitive impairment with or without functional impairment. J Geriatr Psychiatry Neurol. 2012 Dec;25(4):227-32. doi: 10.1177/0891988712464822. Epub 2012 Nov 21. PMID 23172761
- [Result] Song J, Wang S, Tan M, Jia J. G1/S checkpoint proteins in peripheral blood lymphocytes are potentially diagnostic biomarkers for Alzheimer's disease. Neurosci Lett. 2012 Sep 27;526(2):144-9. doi: 10.1016/j.neulet.2012.08.020. Epub 2012 Aug 17. PMID 22922216
- [Result] Tan M, Wang S, Song J, Jia J. Combination of p53(ser15) and p21/p21(thr145) in peripheral blood lymphocytes as potential Alzheimer's disease biomarkers. Neurosci Lett. 2012 May 16;516(2):226-31. doi: 10.1016/j.neulet.2012.03.093. Epub 2012 Apr 6. PMID 22503900
- [Result] Wang F, Shu C, Jia L, Zuo X, Zhang Y, Zhou A, Qin W, Song H, Wei C, Zhang F, Hong Z, Tang M, Wang DM, Jia J. Exploration of 16 candidate genes identifies the association of IDE with Alzheimer's disease in Han Chinese. Neurobiol Aging. 2012 May;33(5):1014.e1-9. doi: 10.1016/j.neurobiolaging.2010.08.004. Epub 2010 Sep 28. PMID 20880607
- [Result] Wang S, Song J, Tan M, Albers KM, Jia J. Mitochondrial fission proteins in peripheral blood lymphocytes are potential biomarkers for Alzheimer's disease. Eur J Neurol. 2012 Jul;19(7):1015-22. doi: 10.1111/j.1468-1331.2012.03670.x. Epub 2012 Feb 16. PMID 22340708
- [Result] Xing Y, Qin W, Li F, Jia XF, Jia J. Apolipoprotein E epsilon4 status modifies the effects of sex hormones on neuropsychiatric symptoms of Alzheimer's disease. Dement Geriatr Cogn Disord. 2012;33(1):35-42. doi: 10.1159/000336600. Epub 2012 Mar 2. PMID 22398564
- [Result] Xing Y, Wei C, Chu C, Zhou A, Li F, Wu L, Song H, Zuo X, Wang F, Qin W, Li D, Tang Y, Jia XF, Jia J. Stage-specific gender differences in cognitive and neuropsychiatric manifestations of vascular dementia. Am J Alzheimers Dis Other Demen. 2012 Sep;27(6):433-8. doi: 10.1177/1533317512454712. PMID 22930700
- [Result] Li F, Wang F, Jia J. Evaluating the prevalence of dementia in hospitalized older adults and effects of comorbid dementia on patients' hospital course. Aging Clin Exp Res. 2013 Aug;25(4):393-401. doi: 10.1007/s40520-013-0068-z. Epub 2013 Jul 20. PMID 23872925
- [Result] Xing Y, Qin W, Li F, Jia XF, Jia J. Associations between sex hormones and cognitive and neuropsychiatric manifestations in vascular dementia (VaD). Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):85-90. doi: 10.1016/j.archger.2012.10.003. Epub 2012 Oct 24. PMID 23103091
- [Result] Jia J, Wang F, Wei C, Zhou A, Jia X, Li F, Tang M, Chu L, Zhou Y, Zhou C, Cui Y, Wang Q, Wang W, Yin P, Hu N, Zuo X, Song H, Qin W, Wu L, Li D, Jia L, Song J, Han Y, Xing Y, Yang P, Li Y, Qiao Y, Tang Y, Lv J, Dong X. The prevalence of dementia in urban and rural areas of China. Alzheimers Dement. 2014 Jan;10(1):1-9. doi: 10.1016/j.jalz.2013.01.012. Epub 2013 Jul 18. PMID 23871765
- [Result] Jia J, Zhou A, Wei C, Jia X, Wang F, Li F, Wu X, Mok V, Gauthier S, Tang M, Chu L, Zhou Y, Zhou C, Cui Y, Wang Q, Wang W, Yin P, Hu N, Zuo X, Song H, Qin W, Wu L, Li D, Jia L, Song J, Han Y, Xing Y, Yang P, Li Y, Qiao Y, Tang Y, Lv J, Dong X. The prevalence of mild cognitive impairment and its etiological subtypes in elderly Chinese. Alzheimers Dement. 2014 Jul;10(4):439-447. doi: 10.1016/j.jalz.2013.09.008. Epub 2014 Jan 10. PMID 24418053
- [Result] Qin W, Jia X, Wang F, Zuo X, Wu L, Zhou A, Li D, Min B, Wei C, Tang Y, Xing Y, Dong X, Wang Q, Gao Y, Li Y, Jia J. Elevated plasma angiogenesis factors in Alzheimer's disease. J Alzheimers Dis. 2015;45(1):245-52. doi: 10.3233/JAD-142409. PMID 25690662
- [Result] Song H, Long H, Zuo X, Yu C, Liu B, Wang Z, Wang Q, Wang F, Han Y, Jia J. APOE Effects on Default Mode Network in Chinese Cognitive Normal Elderly: Relationship with Clinical Cognitive Performance. PLoS One. 2015 Jul 15;10(7):e0133179. doi: 10.1371/journal.pone.0133179. eCollection 2015. PMID 26177270
- [Result] Jia J, Zuo X, Jia XF, Chu C, Wu L, Zhou A, Wei C, Tang Y, Li D, Qin W, Song H, Ma Q, Li J, Sun Y, Min B, Xue S, Xu E, Yuan Q, Wang M, Huang X, Fan C, Liu J, Ren Y, Jia Q, Wang Q, Jiao L, Xing Y, Wu X; China Cognition and Aging Study (China COAST) Group. Diagnosis and treatment of dementia in neurology outpatient departments of general hospitals in China. Alzheimers Dement. 2016 Apr;12(4):446-53. doi: 10.1016/j.jalz.2015.06.1892. Epub 2015 Aug 7. PMID 26256457
- [Result] Li H, Jia J, Yang Z. Mini-Mental State Examination in Elderly Chinese: A Population-Based Normative Study. J Alzheimers Dis. 2016 May 7;53(2):487-96. doi: 10.3233/JAD-160119. PMID 27163822
- [Result] Xing Y, Tang Y, Zhao L, Wang Q, Qin W, Zhang JL, Jia J. Plasma Ceramides and Neuropsychiatric Symptoms of Alzheimer's Disease. J Alzheimers Dis. 2016 Apr 12;52(3):1029-35. doi: 10.3233/JAD-151158. PMID 27079712
- [Result] Yuan X, Han Y, Wei Y, Xia M, Sheng C, Jia J, He Y. Regional homogeneity changes in amnestic mild cognitive impairment patients. Neurosci Lett. 2016 Aug 26;629:1-8. doi: 10.1016/j.neulet.2016.06.047. Epub 2016 Jun 23. PMID 27345927
- [Result] Li D, Hu N, Yu Y, Zhou A, Li F, Jia J. Trajectories of Multidimensional Caregiver Burden in Chinese Informal Caregivers for Dementia: Evidence from Exploratory and Confirmatory Factor Analysis of the Zarit Burden Interview. J Alzheimers Dis. 2017;59(4):1317-1325. doi: 10.3233/JAD-170172. PMID 28759966
- [Result] Liu Q, Zhu Z, Teipel SJ, Yang J, Xing Y, Tang Y, Jia J. White Matter Damage in the Cholinergic System Contributes to Cognitive Impairment in Subcortical Vascular Cognitive Impairment, No Dementia. Front Aging Neurosci. 2017 Feb 27;9:47. doi: 10.3389/fnagi.2017.00047. eCollection 2017. PMID 28289381
- [Result] Jia J, Wei C, Chen S, Li F, Tang Y, Qin W, Zhao L, Jin H, Xu H, Wang F, Zhou A, Zuo X, Wu L, Han Y, Han Y, Huang L, Wang Q, Li D, Chu C, Shi L, Gong M, Du Y, Zhang J, Zhang J, Zhou C, Lv J, Lv Y, Xie H, Ji Y, Li F, Yu E, Luo B, Wang Y, Yang S, Qu Q, Guo Q, Liang F, Zhang J, Tan L, Shen L, Zhang K, Zhang J, Peng D, Tang M, Lv P, Fang B, Chu L, Jia L, Gauthier S. The cost of Alzheimer's disease in China and re-estimation of costs worldwide. Alzheimers Dement. 2018 Apr;14(4):483-491. doi: 10.1016/j.jalz.2017.12.006. Epub 2018 Feb 9. PMID 29433981
- [Result] Li J, Wu L, Tang Y, Zhou A, Wang F, Xing Y, Jia J. Differentiation of neuropsychological features between posterior cortical atrophy and early onset Alzheimer's disease. BMC Neurol. 2018 May 10;18(1):65. doi: 10.1186/s12883-018-1068-6. PMID 29747584
- [Result] Qiu Q, Shen L, Jia L, Wang Q, Li F, Li Y, Jia J. A Novel PSEN1 M139L Mutation Found in a Chinese Pedigree with Early-Onset Alzheimer's Disease Increases Abeta42/Abeta40 ratio. J Alzheimers Dis. 2019;69(1):199-212. doi: 10.3233/JAD-181291. PMID 30958370
- [Result] Jia L, Qiu Q, Zhang H, Chu L, Du Y, Zhang J, Zhou C, Liang F, Shi S, Wang S, Qin W, Wang Q, Li F, Wang Q, Li Y, Shen L, Wei Y, Jia J. Concordance between the assessment of Abeta42, T-tau, and P-T181-tau in peripheral blood neuronal-derived exosomes and cerebrospinal fluid. Alzheimers Dement. 2019 Aug;15(8):1071-1080. doi: 10.1016/j.jalz.2019.05.002. PMID 31422798
- [Result] Jia L, Fu Y, Shen L, Zhang H, Zhu M, Qiu Q, Wang Q, Yan X, Kong C, Hao J, Wei C, Tang Y, Qin W, Li Y, Wang F, Guo D, Zhou A, Zuo X, Yu Y, Li D, Zhao L, Jin H, Jia J. PSEN1, PSEN2, and APP mutations in 404 Chinese pedigrees with familial Alzheimer's disease. Alzheimers Dement. 2020 Jan;16(1):178-191. doi: 10.1002/alz.12005. PMID 31914229
- [Result] Zhao T, Quan M, Jia J. Functional Connectivity of Default Mode Network Subsystems in the Presymptomatic Stage of Autosomal Dominant Alzheimer's Disease. J Alzheimers Dis. 2020;73(4):1435-1444. doi: 10.3233/JAD-191065. PMID 31929167
- [Result] Quan M, Zhao T, Tang Y, Luo P, Wang W, Qin Q, Li T, Wang Q, Fang J, Jia J. Effects of gene mutation and disease progression on representative neural circuits in familial Alzheimer's disease. Alzheimers Res Ther. 2020 Jan 14;12(1):14. doi: 10.1186/s13195-019-0572-2. PMID 31937364
- [Result] Jia L, Xu H, Chen S, Wang X, Yang J, Gong M, Wei C, Tang Y, Qu Q, Chu L, Shen L, Zhou C, Wang Q, Zhao T, Zhou A, Li Y, Li F, Li Y, Jin H, Qin Q, Jiao H, Li Y, Zhang H, Lyu D, Shi Y, Song Y, Jia J. The APOE epsilon4 exerts differential effects on familial and other subtypes of Alzheimer's disease. Alzheimers Dement. 2020 Dec;16(12):1613-1623. doi: 10.1002/alz.12153. Epub 2020 Sep 3. PMID 32881347
- [Result] Jia L, Zhu M, Kong C, Pang Y, Zhang H, Qiu Q, Wei C, Tang Y, Wang Q, Li Y, Li T, Li F, Wang Q, Li Y, Wei Y, Jia J. Blood neuro-exosomal synaptic proteins predict Alzheimer's disease at the asymptomatic stage. Alzheimers Dement. 2021 Jan;17(1):49-60. doi: 10.1002/alz.12166. Epub 2020 Aug 10. PMID 32776690
- [Result] Han Y, Zhou A, Li F, Wang Q, Xu L, Jia J. Apolipoprotein E epsilon4 allele is associated with vascular cognitive impairment no dementia in Chinese population. J Neurol Sci. 2020 Feb 15;409:116606. doi: 10.1016/j.jns.2019.116606. Epub 2019 Dec 6. PMID 31865187
- [Result] Qiu Q, Jia L, Wang Q, Zhao L, Jin H, Li T, Quan M, Xu L, Li B, Li Y, Jia J. Identification of a novel PSEN1 Gly111Val missense mutation in a Chinese pedigree with early-onset Alzheimer's disease. Neurobiol Aging. 2020 Jan;85:155.e1-155.e4. doi: 10.1016/j.neurobiolaging.2019.05.018. Epub 2019 May 31. PMID 31235344
- [Result] Jia L, Du Y, Chu L, Zhang Z, Li F, Lyu D, Li Y, Li Y, Zhu M, Jiao H, Song Y, Shi Y, Zhang H, Gong M, Wei C, Tang Y, Fang B, Guo D, Wang F, Zhou A, Chu C, Zuo X, Yu Y, Yuan Q, Wang W, Li F, Shi S, Yang H, Zhou C, Liao Z, Lv Y, Li Y, Kan M, Zhao H, Wang S, Yang S, Li H, Liu Z, Wang Q, Qin W, Jia J; COAST Group. Prevalence, risk factors, and management of dementia and mild cognitive impairment in adults aged 60 years or older in China: a cross-sectional study. Lancet Public Health. 2020 Dec;5(12):e661-e671. doi: 10.1016/S2468-2667(20)30185-7. PMID 33271079
- [Result] Jia L, Li F, Wei C, Zhu M, Qu Q, Qin W, Tang Y, Shen L, Wang Y, Shen L, Li H, Peng D, Tan L, Luo B, Guo Q, Tang M, Du Y, Zhang J, Zhang J, Lyu J, Li Y, Zhou A, Wang F, Chu C, Song H, Wu L, Zuo X, Han Y, Liang J, Wang Q, Jin H, Wang W, Lu Y, Li F, Zhou Y, Zhang W, Liao Z, Qiu Q, Li Y, Kong C, Li Y, Jiao H, Lu J, Jia J. Prediction of Alzheimer's disease using multi-variants from a Chinese genome-wide association study. Brain. 2021 Apr 12;144(3):924-937. doi: 10.1093/brain/awaa364. PMID 33188687
- [Result] Qin W, Zhou A, Zuo X, Jia L, Li F, Wang Q, Li Y, Wei Y, Jin H, Cruchaga C, Benitez BA, Jia J. Exome sequencing revealed PDE11A as a novel candidate gene for early-onset Alzheimer's disease. Hum Mol Genet. 2021 May 28;30(9):811-822. doi: 10.1093/hmg/ddab090. PMID 33835157
- [Result] Jia J, Zhao T, Liu Z, Liang Y, Li F, Li Y, Liu W, Li F, Shi S, Zhou C, Yang H, Liao Z, Li Y, Zhao H, Zhang J, Zhang K, Kan M, Yang S, Li H, Liu Z, Ma R, Lv J, Wang Y, Yan X, Liang F, Yuan X, Zhang J, Gauthier S, Cummings J. Association between healthy lifestyle and memory decline in older adults: 10 year, population based, prospective cohort study. BMJ. 2023 Jan 25;380:e072691. doi: 10.1136/bmj-2022-072691. PMID 36696990
- [Result] Jia J, Zhang Y, Shi Y, Yin X, Wang S, Li Y, Zhao T, Liu W, Zhou A, Jia L. A 19-Year-Old Adolescent with Probable Alzheimer's Disease. J Alzheimers Dis. 2023;91(3):915-922. doi: 10.3233/JAD-221065. PMID 36565128
- [Result] Li W, Pang Y, Wang Y, Mei F, Guo M, Wei Y, Li X, Qin W, Wang W, Jia L, Jia J. Aberrant palmitoylation caused by a ZDHHC21 mutation contributes to pathophysiology of Alzheimer's disease. BMC Med. 2023 Jun 26;21(1):223. doi: 10.1186/s12916-023-02930-7. PMID 37365538
- [Result] Quan M, Wang Q, Qin W, Wang W, Li F, Zhao T, Li T, Qiu Q, Cao S, Wang S, Wang Y, Jin H, Zhou A, Fang J, Jia L, Jia J. Shared and unique effects of ApoEepsilon4 and pathogenic gene mutation on cognition and imaging in preclinical familial Alzheimer's disease. Alzheimers Res Ther. 2023 Feb 28;15(1):40. doi: 10.1186/s13195-023-01192-y. PMID 36850008
- [Result] Jia J, Ning Y, Chen M, Wang S, Yang H, Li F, Ding J, Li Y, Zhao B, Lyu J, Yang S, Yan X, Wang Y, Qin W, Wang Q, Li Y, Zhang J, Liang F, Liao Z, Wang S. Biomarker Changes during 20 Years Preceding Alzheimer's Disease. N Engl J Med. 2024 Feb 22;390(8):712-722. doi: 10.1056/NEJMoa2310168. PMID 38381674
- [Derived] Zhao B, Zang P, Quan M, Wang Q, Guo D, Jia J, Wang W. The Effect of APOE epsilon4 on Alzheimer's Disease Fluid Biomarkers: A Cross-Sectional Study Based on the COAST. CNS Neurosci Ther. 2025 Jan;31(1):e70202. doi: 10.1111/cns.70202. PMID 39749650
- See also: COAST Website — http://ad.chinacfan.org/Default.aspx

DOCUMENTS (1):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT03653156/Prot_000.pdf